CLINICAL TRIAL: NCT04613271
Title: Phase III, Random-Open, Clinical Trials on the Efficacy and Safety of Favipiravir in Covid-19 Patients in Indonesia
Brief Title: Efficacy and Safety of Favipiravir in Covid-19 Patients in Indonesia
Acronym: FVR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ina-Respond (Other)
Collaborators: Center for Research and Development of Health Resources and Services, National Institute of Health Research and Development (NIHRD), Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVR; U1111-1263-1797 (Other: WHO UTN Number)
Record Dates: First submitted 2020-10-25; First posted 2020-11-03 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Infectious Disease; SARS-CoV Infection; Covid19
Keywords: Favipiravir; Covid19; SARS-Cov2
MeSH Terms: conditions — Communicable Diseases; Severe Acute Respiratory Syndrome; COVID-19 | interventions — favipiravir; Azithromycin

STUDY DESIGN:
Intervention Model Description: * Group 1: Favipiravir 1600 mg twice a day at day 1 and 600 mg twice a day at day 7-14 + Azithromycin 500 mg once a day for 5 days.
  * Group 2: Azithromycin 500 mg once a day for 5 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Assignment of Administration Group 1:
  Favipiravir 1600 mg twice a day at day 1 and 600 mg twice a day at day 7-14 + Azithromycin 500 mg once a day for 5 days.
  Interventions: Drug: Favipiravir
- Group 2 (Active Comparator): Administration Group 2: Azithromycin 500 mg once a day for 5 days.
  Interventions: Drug: Favipiravir; Drug: Azithromycin

INTERVENTIONS:
Drug: Favipiravir — Assignment of Administration Group 1:
  Favipiravir 1600 mg twice a day at day 1 and 600 mg twice a day at day 7-14 + Azithromycin 500 mg once a day for 5 days.
  Other Names: Treatment Group
Drug: Azithromycin — Azithromycin 500 mg once a day for 5 days.
  Other Names: Group 2
  Arms: Group 2

SUMMARY:
The benefit of the research is to provide information regarding the efficacy and safety of Favipiravir plus the Standard of Care (SoC) for mild-moderate COVID-19 patients to be a reference for policy recommendations regarding the use of Favipiravir as an antiviral drug for the treatment of Covid-19.

DETAILED DESCRIPTION:
Pre-screening is assessing patients who meet the inclusion and exclusion criteria. Screening was carried out to assess whether the subjects met the inclusion and exclusion criteria. Randomization was performed to determine the study drug allocation. The research subjects were inpatients at selected hospitals and at the time of recruitment, the time was called D1. The next day is called D2 and so on Follow-up will be carried out from the first day of recruitment, taking medication up to a maximum of 19 days for test drugs and 11 days for SoC drugs. Recording of clinical and laboratory manifestations will be carried out from recruitment until the patient returns from the hospital.

All results will be recorded in a case report form, and if a case of clinical and laboratory manifestations is found to be severe, it will be written on the adverse case report form and reported immediately according to standard GCP procedures. Subjects may also drop out of the study due to discontinuation of follow-up or a protocol violation

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years - 59 years
2. Confirmation of Covid-19 based on the results of the Real Time PCR (RTPCR) examination for SARS-COV-2 less than 7 days before the first day of taking the drug
3. Patients with mild-moderate clinical manifestations were admitted to the hospital designated by the physician according to the operational definition of the study protocol
4. Have not received COVID-19 antiviral therapy
5. Consciously and voluntarily participate in research

Exclusion Criteria:

1. Pregnant and lactating women
2. Allergy history to Favipiravir and standard hospital drugs
3. Patients with uric acid examination values above normal male> 7 mg / dL; women> 5.7 mg / dL
4. Patients with a history of prolonged ECG / Arrhythmia / QT disorders
5. Cannot swallow drug

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Clinical improvement measured by no sign & symptom for 3 days and RTPCR negative | until 3 days
  Clinical improvement measured by no sign & symptom and RTPCR negative from baseline to Day 3

SECONDARY OUTCOMES:
Duration of hospitalization | until 19 days
  Duration of hospitalization is defined as the number of days in the hospital until Day 19, and descriptive statistics (number of subjects, mean, standard deviation, median, minimum, maximum) are given for each administration group.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. dr. Armedy Ronny Hasugiana, M. Biomed, MD, Principal Investigator — Center for R & D of Health Resources and Services, National Institute of Health Research and Development (NIHRD), Indonesia
Locations (3):
- Indonesia (3):
  - RSJ Soerodjo, Magelang, Central Java
  - RSUP Dr. Kariadi, Semarang, Central of Java
  - RSPI Sulianti Saroso, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No